CLINICAL TRIAL: NCT01037374
Title: Anticipation of the Difficult Airway: the Preoperative Airway Assessment Form as an Educational and Quality Improvement Tool
Brief Title: Anticipation of the Difficult Airway: the Preoperative Airway Assessment Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-0144
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Endotracheal Intubation Risk Assessment
Keywords: risk; assessment; difficult; endotracheal; intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Difficult Airway Assessment Form (Experimental)
  Interventions: Other: Preoperative assessment form

INTERVENTIONS:
Other: Preoperative assessment form — (based on the american society of anesthesiologists)components of the form include: neck measurements; neck mobility; mallampati; wilson's test; pre-existing conditions; and predictions of difficult mask ventilation, supraglottic airway, laryngoscopy, intubation, and surgical airway.

SUMMARY:
The purpose of this study is to see if our experimental preoperative airway assessment form is a better indicator of difficult airway as compared to the anesthesia record that is presently used.

DETAILED DESCRIPTION:
Predicting difficult airway continues to be problematic for even the most seasoned of anesthesiologists. In our study, the resident class will be our sample population. The residents will be randomly assigned into two groups: the experimental group will be utilizing the new preoperative airway assessment form and the control group will be utilizing the standard anesthesia record. Simultaneously, a subset of our anesthesia experts will also be assessing patients preoperatively. The five areas of difficult airway management will be considered: difficult mask ventilation, difficult supraglottic airway, difficult laryngoscopy, difficult intubation, and difficult surgical airway.

According to the American Society of Anesthesiologists, the incidence of intubation has remained stable throughout the 1980s and 1990s despite attempts to predict its occurrence. Many of these cases were considered to be preventable; therefore, a better prediction of and preparation for difficult airway management may lead to a reduction in adverse events.

ELIGIBILITY:
Inclusion Criteria:

* CA-1, CA-2, and CA-3 anesthesiology residents starting from July 2008-July 2010

Exclusion Criteria:

* the same anesthesiology residents who are working with patients 17 and younger, patients who are already intubated, and patients undergoing emergent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Use of an experimental preoperative assessment form by residents will result in more complete documentation of important airway features compared to use of the current forms | interim analysis will be assessed after 1 year

SECONDARY OUTCOMES:
use of the experimental preoperative assessment form will result in greater resident recognition of patients at high risk for a difficult airway as judged independently by one of 3 senior faculty investigators. | interim analyses will be assessed after 1 year
the percentage of patients intubated using an awake method will be greater among residents using the new form than those using the current form | interim analysis will be assessed after 1 year
the percentage of patients requiring multiple intubation attempts or use of invasive airway techniques will be lower among residents using the new form. | interim analysis will be assessed after 1 year
spontaneous knowledge of important airway features will be more complete among residents using the new form at 18 months of training. | interim analysis will be assessed after 1 year
observations made during this study will allow refinement of the new form to augment the identification of patients with difficult airway. | interim analysis will be assessed after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, MD, Principal Investigator — University of Texas at Houston Health Science Center, Medical School
Locations (1):
- Memorial Hermann Hospital, Medical Center, Houston, Texas, United States

REFERENCES:
- See also: university of texas at houston home page — http://www.uthouston.edu